CLINICAL TRIAL: NCT06786247
Title: Evaluation of an Asynchronous Remote Communities Approach to Behavioral Activation for Depressed Adolescents
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Jessica Jenness, Associate Professor: Department of Psychiatry and Behavioral Sciences, University of Washington
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00018887; 5R34MH128387-02 (NIH)
Record Dates: First submitted 2024-12-20; First posted 2025-01-22 (Actual); Last update posted 2025-01-22 (Actual); Status verified 2025-01

CONDITIONS: Depression; Adolescent Behavior
Keywords: depression; adolescence; asynchronous remote community; behavioral activation; digital health
MeSH Terms: conditions — Depression; Adolescent Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ActivaTeen + BA (Experimental): Receives access to ActivaTeen app along with individual behavioral activation therapy
  Interventions: Behavioral: ActivaTeen; Behavioral: Behavioral Activation
- BA Only (Active Comparator): Receives individual behavioral activation therapy alone
  Interventions: Behavioral: Behavioral Activation

INTERVENTIONS:
Behavioral: ActivaTeen — The ActivaTeen app is built on HIPAA-compliant instance of a popular messaging software. Participants in the treatment group can access the app at any time via desktop or mobile, where they can find features designed to enhance their receipt of BA therapy.
  These features include: weekly BA skills and homework completion support, in-app messaging with their BA therapist, mood and activity tracking and data visualizations, chatbot check-ins on progress and guided problem-solving around barriers, and moderated peer support using the ActivaTeen app. The app will have a moderator, who is part of the study team, to manage peer-to-peer interactions within ActivaTeen.
  Arms: ActivaTeen + BA
Behavioral: Behavioral Activation — Behavioral activation therapy involves individual weekly sessions with a trained therapist for 12 weeks. The sessions are completed either in-person or via telehealth. The treatment focuses on behavioral manifestations of depression such as isolating, and how these behaviors are interconnected with low mood and depressive emotions. BA helps patients find ways to engage in behaviors that are meaningful to them based on their values, priorities, and goals, with the aim of creating positive loops between doing meaningful activities and improved mood. The therapist provides structure and problem-solving for activating these behaviors and keeping track of changes over time.
  Other Names: BA

SUMMARY:
The goal of this clinical trial is to learn if a digital health intervention, called "ActivaTeen," improves depression treatment for teenagers with depression. The investigators also want to know if ActivaTeen is easy to use for both teenagers and mental health clinicians who help deliver treatment through ActivaTeen. All teenagers in the study will receive an individual depression therapy called Behavioral Activation or "BA" and about half will also use ActivaTeen.

The main questions this trial aims to answer are:

* Does ActivaTeen improve depression treatment for teenagers?
* Do teenagers and clinicians find ActivaTeen to be acceptable?

Researchers will compare teenagers using ActivaTeen along with BA to teenagers who are only doing BA to see the effects of ActivaTeen.

Participants in the study will:

* Fill out surveys online several times during the study, which lasts about 6 months
* Receive individual BA therapy

ELIGIBILITY:
Inclusion Criteria:

* Age 13 - 19
* Referred for MDD treatment
* Clinically assessed diagnosis of current MDD based on caregiver or patient report or a PHQ-8 total of 8 or greater (moderate MDD)
* MDD clinically determined to be the primary diagnosis
* English-speaking
* Access to a smartphone device

Exclusion Criteria:

* Developmental disability (e.g., intellectual disability, autism spectrum disorder)
* Severe psychiatric comorbidity (e.g., active suicidality requiring higher level of care; psychosis or substance use, bipolar, or conduct disorder)
* Previously completed a full course of evidence based psychosocial intervention for depression

Ages: 13 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 70 (Estimated)
Dates: Start 2025-04 (Estimated); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Intervention Usability Scale | Week 12
  The IUS was adapted from the System Usability Scale, with the word "system" replaced with "intervention platform" for each item. Items are rated on a Likert-type scale from 0 (strongly disagree) to 4 (strongly agree) and half of the items are reverse-scored. The total score is calculated by multiplying the sum of these scores by 2.5 (possible range: 0-100), with higher scores indicating greater usability.
User Burden Scale | Week 12
  The User Burden Scale (UBS) is a widely used and reliable scale that includes 20-items that capture user burden of computing systems across 6 subscales1) difficulty of use, 2) physical, 3) time and social, 4) mental and emotional, 5) privacy, and 6) financial. Items are rated on a 5-point Likert scale from 0 (Never/Not at all) to 4 (All of the time/Extremely). Higher scale scores indicate greater user burden.
Client Satisfaction Questionnaire - 8 | Week 12
  The CSQ-8 is an 8-item, unidimensional measure assessing general satisfaction with mental health services. Higher scores indicate greater satisfaction (range: 8 - 32)
Acceptability Of Intervention Measure | Week 12
  The Acceptability of Intervention Measure assesses the acceptability of a particular intervention. The measure has 4 items each and responses are coded on a 1 - 5 Likert scale (Completely Disagree to Completely Agree). Higher scores indicate greater acceptability (range: 4 - 20)
Intervention Appropriateness Measure | Week 12
  The Intervention Appropriateness Measure assesses the appropriateness of a particular intervention. The measure has 4 items each and responses are coded on a 1 - 5 Likert scale (Completely Disagree to Completely Agree). Higher scores indicate greater appropriateness (range: 4 - 20)
Feasibility Of Intervention Measure | Week 12
  The Feasibility of Intervention Measure assesses the feasibility of a particular intervention. The measure has 4 items each and responses are coded on a 1 - 5 Likert scale (Completely Disagree to Completely Agree). Higher scores indicate greater feasibility (range: 4 - 20)

SECONDARY OUTCOMES:
Loneliness | Baseline to Week 24
  The self-report NIH Loneliness Toolbox assesses perceptions of loneliness in the past month using a 7-item survey for ages 8 to 17 scored on a 5-point Likert scale from 1 (Never) to 5 (Always). Higher total scores indicate greater loneliness. Age-adjusted scale scores will be generated for each participant.
Therapeutic Alliance | Week 12
  The Working Alliance Inventory, Short Form (WAI-S) will be used to assess the therapeutic alliance between clients and therapists. The WAI-S comprises 12 items designed to evaluate the quality of the working relationship, agreement on goals, and agreement on tasks between the client and therapist. Each item is scored on a 1 to 7 Likert scale, where higher scores indicate stronger therapeutic alliance. The total score ranges from 12 to 84, with higher scores indicating a more positive and effective therapeutic alliance.

OTHER OUTCOMES:
Enrollment Rate | Baseline
  The enrollment rate (those enrolled / those screened) will be used as a measure of trial design feasibility. The number of participants enrolled will be divided by the number of candidates screened.
Loss to Follow Up Rate | Baseline to Week 24
  The loss-to-follow-up rate (participants who do not complete Week 24 / randomized participants) will be used as a measure of trial design feasibility. The number of participants who do not complete the Week 24 visit will be divided by the number of participants who complete randomization.
Behavioral Activation Attendance | Baseline to Week 12
  Attendance at BA sessions will be used as a measure of engagement in treatment (both study arms receive BA). The number of attended sessions will be divided by the total possible (12).
Behavioral Activation Homework Completion | Baseline to Week 12
  Completion of BA homework will be used as a measure of engagement in treatment (both study arms receive BA). The number of completed homeworks will be divided by the total possible.
Behavioral Activation Skill Use | Baseline to Week 12
  This weekly checklist measures whether or not BA skills are used outside of session. BA skills include Goal Directed Behavior, Tracking Mood-Activities, Mood Boosting Activities, SMART Goal setting, Mini-step Completion, Problem-solving, Making the Most of a Good Moment. The number of skills completed per week will be summed (range: 0 -7) and averaged across the study period. Higher scores indicate greater BA skill use.
ActivaTeen - Time Spent on Platform | Baseline to Week 12
  The amount of time spent on the intervention platform (ActivaTeen) will be measured and recorded. We will use a cut off of XX mins per day as a threshold for low engagement.
ActivaTeen - Messaging Rates | Baseline to Week 12
  Frequency of direct messages sent to other teens and to their assigned clinician via the general Teams chat and/or ActivaTeen Team chat.
Treatment-Related Adverse Events | Baseline to Week 24
  Intervention safety will be assessed by comparing the number of adverse events per person that are "definitely" or "probably" attributable to study procedures across treatment arms.
Suicidality | Baseline to Week 24
  Suicidality will be assessed with 4 items from the Mood and Feelings Questionnaire (MFQ) called the MFQ-SI (for Suicidal Ideation). Items are rated on a 1 - 3 Likert Scale (Not True, Sometimes, True) and summed with higher total scores indicating greater suicidality.
Depression Symptoms | Baseline to Week 24
  Symptoms of depression will be measured with the 9-item Patient Health Questionnaire (PHQ-9). The PHQ-9 consists of nine questions based on the criteria for major depressive disorder in the DSM-5.Each question is scored on a 0 - 3 Likert scale, with 0 representing "not at all" and 3 representing "nearly every day." The total score ranges from 0 to 27, with higher scores indicating more severe depressive symptoms.
Anxiety Symptoms | Baseline to Week 24
  Symptoms of generalized anxiety disorder (GAD) will be assessed using the 7-item Generalized Anxiety Disorder scale (GAD-7). The GAD-7 comprises seven questions designed to evaluate the severity of anxiety symptoms based on criteria in the DSM-5. Each question is rated on a 0 to 3 Likert scale, where 0 indicates "not at all" and 3 indicates "nearly every day." The total score on the GAD-7 ranges from 0 to 21, with higher scores indicating greater anxiety symptoms.
Major Depressive Disorder | Baseline to Week 24
  The Children's Depression Rating Scale-Revised (CDRS-R) will be utilized to assess depression symptoms in children and adolescents. The CDRS-R is a clinician-rated scale comprising 17 items that evaluate various aspects of depression, such as mood, behavior, and physical symptoms. Each item is scored on a scale from 1 to 5, with higher scores indicating more severe depressive symptoms. The total score ranges from 17 to 85, with higher scores indicating greater depression severity.
Externalizing psychopathology symptoms | Baseline to Week 24
  The Strengths and Difficulties Questionnaire (SDQ) will be used to assess various aspects of children's emotional and behavioral functioning. The SDQ consists of 25 items that cover emotional symptoms, conduct problems, hyperactivity/inattention, peer relationship problems, and prosocial behavior. Each item is rated on a 3-point scale (0 = not true, 1 = somewhat true, 2 = certainly true). Subscale scores are generated for emotional symptoms, conduct problems, hyperactivity/inattention, peer relationship problems, and prosocial behavior. Higher scores indicate higher levels of emotional and behavioral difficulties.
Client-Centeredness of Treatment | Week 12
  The Giving Youth a Voice Short Form questionnaire (GYVSF) will be utilized to assess participant perspectives on the treatment they received in the study. The GYV-SF includes items designed to capture youths' opinions on topics such as education, relationships, and community engagement. Each item is rated on a 7-point Likert scale with higher scores indicating perceptions of more client-centered behaviors from service providers.

CONTACTS AND LOCATIONS:
Overall Officials: Jessica Jenness, PhD, Principal Investigator — University of Washington

DOCUMENTS (3):
  • Study Protocol (2024-01-29): https://cdn.clinicaltrials.gov/large-docs/47/NCT06786247/Prot_000.pdf
  • Statistical Analysis Plan (2024-01-29): https://cdn.clinicaltrials.gov/large-docs/47/NCT06786247/SAP_001.pdf
  • Informed Consent Form (2024-01-29): https://cdn.clinicaltrials.gov/large-docs/47/NCT06786247/ICF_002.pdf